CLINICAL TRIAL: NCT01867684
Title: Brief Positive Psychotherapy After Acquired Brain Injury: A Pilot Randomised Controlled Trial
Brief Title: Positive PsychoTherapy in Acquired Brain Injury (ABI) Rehabilitation
Acronym: PoPsTAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GN12CP391; CZH/4/778 (Other Grant/Funding Number: Chief Scientist Office)
Record Dates: First submitted 2013-05-20; First posted 2013-06-04 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Acquired Brain Injury; Emotional Distress
Keywords: Stroke; Acquired brain injury
MeSH Terms: conditions — Brain Injuries; Stroke | interventions — Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment as usual (No Intervention): Standard NHS care for the patient group (NHS care will vary as participants will be recruited from a variety of NHS clinics).
- Psychotherapy (Experimental): Brief psychotherapy intervention delivered over 8 weeks in addition to standard care.
  Interventions: Other: Psychotherapy

INTERVENTIONS:
Other: Psychotherapy
  Arms: Psychotherapy

SUMMARY:
Stroke, head injury and other forms of brain injury are a major cause of physical, psychological and social disability in the adult population. Psychological distress is common following brain injury, but the evidence base for specific psychotherapeutic methods in this population is limited, and standard treatment approaches may not be suitable. Recently there has been a growing interest in positive psychology - the study of wellbeing, positive emotions and characteristics, and personal growth. The investigators believe that positive psychotherapy interventions may be beneficial after acquired brain injury, to reduce psychological morbidity. Because such interventions have not previously been applied in this population, the investigators propose to conduct a pilot randomised controlled trial to examine the feasibility of a brief positive psychotherapy intervention in an out-patient setting. This project will produce essential information to allow us to plan future full-scale clinical trials in this area.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over;
* Diagnosis of stroke or acquired brain injury (confirmed clinically and/or radiologically);
* Between 3 and 12 months post-injury at time of recruitment;
* Presence of emotional distress (score in moderate or above range on at least one sub-scale of the Depression Anxiety Stress Scales; DASS-21);
* Medically stable;
* Able to consent to research.

Exclusion Criteria:

* Significant communication impairments that would preclude participation;
* Diagnosis of mild traumatic brain injury (due to the known additional complexities contributing to outcome in this population);
* Comorbid developmental learning disability or degenerative neurological condition.

Pre-injury history of mood disorder will not lead to exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-07; Primary Completion 2014-05 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Recruitment rate at 20 weeks from baseline | 20 weeks
Treatment adherence at 20 weeks from baseline | 20 weeks
Sample retention at 20 weeks from baseline | 20 weeks

SECONDARY OUTCOMES:
Correlation coefficient between first and second baseline administrations of the Authentic Happiness Inventory (AHI) and VIA-IS questionnaires | 1 week
Change in Depression Anxiety Stress Scales (DASS-21) scores at 20 weeks from baseline | 20 weeks
Changes in AHI scores at 20 weeks from baseline | 20 weeks
Likert ratings of participants and therapists experiences of treatment delivery | 8 weeks
Changes in Mayo-Portland Adaptability Inventory (MPAI-4) scores at 20 weeks at baseline | 20 weeks
Changes in Modified Caregiver Strain Index (MCSI) scores at 20 weeks from baseline | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Evans, PhD, Principal Investigator — University of Glasgow
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom